CLINICAL TRIAL: NCT01469663
Title: Event Related Potentials in Borderline Personality Disorder and Major Depression
Status: Terminated | Type: Observational
Why Stopped: software problem
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Syracuse University (Other)
Responsible Party: Principal Investigator, Amruther G Ramamurthy, Assistant Professor, Dept of Psychiatry, State University of New York - Upstate Medical University
Other Study IDs: 5910
Record Dates: First submitted 2010-10-26; First posted 2011-11-10 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Borderline Personality Disorder; Major Depression
Keywords: Borderline Personality Disorder; Major Depression; Electroencephalogram; N2; Error Related Negativity; Emotional Processing; Levels of Emotional Awareness
MeSH Terms: conditions — Borderline Personality Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy Control: Healthy participants without borderline personality or depression
- Major Depression, No Borderline Personality Disorder: With major depression and no borderline personality
- Major Depression + Borderline Personality Disorder: With major depression and borderline personality disorder
- No Major Depression, Borderline Personality Disorder: With no major depression, but with borderline personality disorder

SUMMARY:
This study examines whether depression in people with borderline personality disorder is different than depression in people without borderline personality disorder.

Unlike people who have depression alone (i.e. without borderline personality disorder), people with borderline personality disorder have depressions that often do not improve with medications. This makes treating depression much more challenging in someone with borderline personality disorder than without borderline personality disorder.

Borderline personality disorderis associated with difficulty in understanding and communicating feelings. Impaired emotion processing may reflect dysfunction of an area of the brain, the anterior cingulate.

Depression is associated with changes in anterior cingulate activity. The investigators believe that when borderline personality disorder is present with depression, brain activity changes in the anterior cingulate will not be the same as in depressed patients without borderline personality disorder.

An electroencephalogram records brain electrical activity. In this study, the investigators will measure electroencephalogram indices reflecting anterior cingulate activity.

HYPOTHESIS: In this study, the investigators predict that when borderline personality is present with depression, electroencephalogram indices of anterior cingulate activity will be different from when depression is present alone (without borderline personality). This could help to explain why people with borderline personality have depressions that are harder to treat than depressions in people without borderline personality.

The investigators also predict that electroencephalogram indices of the anterior cingulate will reflect emotional processing ability, as measured by validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45
* female
* noncontrols diagnosis: major depression &/or borderline personality disorder
* Control participants should have neither major depression or borderline pers.
* meet Structured Controlled Interview for DSM - II cut off scores
* meet Beck Depression Inventory (BDI)cut off scores
* meet Borderline Evaluation of Severity Over Time(BEST) cut off scores.

Exclusion Criteria:

* based on having none of the below diagnoses from patient history, prior clinical records and based on MINI Plus International Neuropsychiatry Interview
* schizophrenia
* psychosis
* Attention Deficit Hyperactivity Disorder
* Obsessive Compulsive Disorder
* bipolar disorder
* mental retardation
* dementia
* CNS disease
* Post-Traumatic Stress Disorder in non-borderline personality disorder groups
* Recreational drug or alcohol use in the past week.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females between age 18 to 45 recruited from staff (healthy controls) or from Upstate Medical University primary care outpatients, psychiatry outpatients, psychiatry inpatients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Error related negativity amplitude | on day 1 and then 4 weeks (average) later
  electroencephalogram amplitude of the error related negativity
N2 amplitude | on day 1 and then 4 weeks (average) later
  electroencephalogram amplitude of N2 wave

CONTACTS AND LOCATIONS:
Overall Officials: Amruthur Ramamurthy, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (2):
- United States (2):
  - Syracuse University - CNY Medical Center, Syracuse, New York
  - Upstate Medical University, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No
There is no useful data